CLINICAL TRIAL: NCT01361334
Title: Phase II Pilot Clinical Trial of Pazopanib in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) or at Initial Diagnosis When no Intensive Treatment is Possible
Brief Title: Pilot Clinical Trial of Pazopanib in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) or at Initial Diagnosis When no Intensive Treatment is Possible
Acronym: PAZOPANIB-AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM09_0018_PAZOPANIB_AML 2011; 2010-024526-37 (EudraCT Number)
Record Dates: First submitted 2011-05-17; First posted 2011-05-26 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2016-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: (other than AML M3)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib (Experimental): Pazopanib treatment
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg QD p.o.
  Other Names: Votrient(R)

SUMMARY:
Long term disease-free survival (DFS) of patients with acute myeloid leukemia (AML) is still poor. Recently, so-called "targeted therapy" for cancer has been introduced to the treatment of patients with AML. This phase II clinical trial will explore the efficacy, safety, and pharmacodynamics of the tyrosine kinase inhibitor pazopanib in patients with relapsed or refractory AML or patients with AML who are not eligible for intensive treatment. Biomarker studies will be included to study whether the targets are indeed inhibited and whether this leads to decreased BM angiogenesis. Toxicity assessments will be included, and the antileukemic effectiveness will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments which are not routinely performed for diagnosis or monitoring of acute myeloid leukemia (AML), and the subjects must be willing to comply with treatment and to follow up assessments and procedures
2. Histologically or cytologically confirmed diagnosis of AML relapsed after or refractory to at least one induction regimen, or patients with AML at initial diagnosis who are not eligible for allogeneic transplant or intensive induction chemotherapy, except for AML M3 (acute promyelocytic leukemia)
3. Age at least 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤3
5. Measurable disease burden (blasts in BM and/or PB, extramedullary blasts [chloroma])
6. Able to swallow and retain oral medication
7. A life expectancy of at least 4 weeks
8. Adequate contraception methods
9. Adequate organ function as defined in the study protocol

Exclusion Criteria:

1. Patients with a valid option for intensive chemotherapy and/or stem cell transplantation (Patients after allogeneic stem cell transplant must be off immunosuppressive agents for at least 2 weeks prior to study entry and Graft-versus host disease must have resolved to Grade ≤2)
2. History of cancer that according to the Investigator might confound the assessment of the endpoints of the study
3. Uncontrolled peptic ulcer disease or clinically significant gastrointestinal abnormalities which interfere with oral dosing or any unstable or serious concurrent condition (e.g., active uncontrolled infection)
4. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥90 mmHg]. Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for the study
5. Prolongation of corrected QT interval (QTc) >480 milliseconds
6. History of any one of more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, symptomatic peripheral vascular disease, class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
7. History of cerebrovascular infarction or bleeding, pulmonary embolism, or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulant agents for at least 6 weeks are eligible
8. Evidence of serious active bleeding or bleeding diathesis (except for bleeding or petechiae due to AML-related thrombocytopenia which will be treated using platelet transfusions). Also, patients with known endobronchial lesions and/or lesions infiltrating major pulmonary vessels will be excluded from the study due to excess risk of bleeding.
9. Prior major surgery or trauma within 28 days prior to first dose of study drug
10. Treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer prior to the first dose of study drug (for bevacizumab 60 days).
11. Concurrent cytoreductive chemotherapy (hydroxyurea must be discontinued at least one day before start of study medication)
12. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to pazopanib
13. Patients with psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
14. Pregnant or lactating and actively breastfeeding patients
15. Patients taking any of the following prohibited medication:

    * clarithromycin, telithromycin, troleandomycin (antibiotics)
    * ritonavir, indinavir, saquinavir, nelfinavir, amprenavir, lopinavir (HIV protease inhibitors)
    * itraconazole, ketoconazole, voriconazole, fluconazole (antifungals)
    * nefazodone (antidepressant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cumulative response rate (CR, CRp, CRi, PR) within up to one year of pazopanib treatment | 12 months
Reduction of BM microvessel density on day 28 | 28 days

SECONDARY OUTCOMES:
Safety and Tolerability (Rate of adverse events) | 12 months
  Rate of adverse events
Cumulative incidence and degree of inhibition of target receptor phosphorylation (PDGFR, VEGFR, and c-KIT) and correlation with clinical response | 12 months
Reduction of BM microvessel density on day 14 | 14 days
Relapse-free survival in relationship to historical control patients, Overall survival in relationship to historical control patients, Duration of response | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Kessler, MD, Principal Investigator — University of Münster, Department of Medicine A, Germany
Locations (1):
- Unviersity Hospital of Münster (UKM), Münster, Germany

REFERENCES:
- [Derived] Kessler T, Koschmieder S, Schliemann C, Crysandt M, Mikesch JH, von Stillfried S, Stelljes M, Pohlen M, Lenz G, Kirsch A, Vehring K, Wardelmann E, Hartmann W, Bormann E, Gerss J, Brummendorf TH, Muller-Tidow C, Berdel WE. Phase II clinical trial of pazopanib in patients with acute myeloid leukemia (AML), relapsed or refractory or at initial diagnosis without an intensive treatment option (PazoAML). Ann Hematol. 2019 Jun;98(6):1393-1401. doi: 10.1007/s00277-019-03651-9. Epub 2019 Mar 21. PMID 30903275